CLINICAL TRIAL: NCT02717611
Title: A Phase 2 Study of the Efficacy and Safety of ACP-196 in Subjects With Relapsed/Refractory CLL and Intolerant of Ibrutinib Therapy
Brief Title: A Study of ACP-196 (Acalabrutinib) in Subjects With Relapsed/Refractory CLL and Intolerant of Ibrutinib Therapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-CL-208; 2015-005317-68 (EudraCT Number)
Record Dates: First submitted 2016-03-11; First posted 2016-03-24 (Estimated); Results first posted 2022-02-09 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Ibrutinib Intolerant
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACP-196 (acalabrutinib) (Experimental): ACP-196 (acalabrutinib) 100 mg to be administered orally (PO) twice a day BID
  Interventions: Drug: ACP-196 (acalabrutinib)

INTERVENTIONS:
Drug: ACP-196 (acalabrutinib) — ACP-196 100 mg to be administered orally (PO) twice a day BID.
  Other Names: Acalabrutinib

SUMMARY:
A Phase 2 Study to evaluate the Efficacy and Safety of ACP-196 (acalabrutinib) in Subjects with Relapsed/Refractory CLL and Intolerant of Ibrutinib Therapy

DETAILED DESCRIPTION:
A Multicenter, Open-Label, Phase 2 study evaluating the efficacy and safety of Acalabrutinib in subjects with relapsed/refractory CLL (N=60) who are intolerant of ibrutinib therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 18 years of age.
2. Prior diagnosis of CLL
3. Must have received ≥ 1 prior therapy for CLL
4. Intolerant of ibrutinib
5. Documented disease progression after stopping ibrutinib therapy as defined by the IWCLL 2008 criteria
6. Willing and able to participate in all required evaluations and procedures in this study protocol including swallowing capsules without difficulty.
7. ECOG performance status of ≤ 2.

Exclusion Criteria:

1. Ongoing AE attributed to ibrutinib therapy
2. Treatment with systemic anticancer therapy for CLL is prohibited between discontinuation of ibrutinib and enrollment on this trial.
3. Prior exposure to a BCL-2 inhibitor (eg, venetoclax/ABT- 199)
4. Prior malignancy (other than CLL), except for adequately treated basal cell or squamous cell skin cancer, in situ cancer, or other cancer from which the subject has been disease free for ≥ 2 years.
5. Significant cardiovascular disease such as uncontrolled or symptomatic untreated arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification, or QTc > 480 msec at screening. Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll on study.
6. Malabsorption syndrome, disease significantly affecting gastrointestinal function, resection of the stomach, extensive small bowel resection that is likely to affect absorption, symptomatic inflammatory bowel disease, partial or complete bowel obstruction, or gastric restrictions and bariatric surgery, such as gastric bypass.
7. Evidence of active Richter's transformation or any evidence of disease progression on ibrutinib therapy or any BTK inhibitor.
8. CNS involvement by CLL or related Richter's transformation.
9. Known history of human immunodeficiency virus (HIV), serologic status reflecting active hepatitis B or C infection, or any uncontrolled active systemic infection.
10. Uncontrolled autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
11. History of stroke or intracranial hemorrhage within 2 months before the first dose of study drug.
12. History of bleeding diathesis.
13. Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
14. Major surgical procedure within 28 days of first dose of study drug.
15. Requires treatment with a strong CYP3A inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-03-08 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2026-06-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Acerta Clinical Trials, Study Director — 1-888-292-9613; acertamc@dlss.com
Locations (22):
- United States (15):
  - Research Site, Tucson, Arizona
  - Research Site, Concord, California
  - Research Site, La Jolla, California
  - Research Site, Palo Alto, California
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Chicago, Illinois
  - Research Site, Lake Success, New York
  - Research Site, New York, New York
  - Research Site, Columbus, Ohio
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Sherman, Texas
  - Research Site, Seattle, Washington
  - Research Site, Spokane, Washington
  - Research Site, Milwaukee, Wisconsin
- Research Site, Bruges, Belgium
- Research Site, Bordeaux, France
- Research Site, Haifa, Israel
- Research Site, Madrid, Spain
- United Kingdom (3):
  - Research Site, Bournemouth
  - Research Site, Leeds
  - Research Site, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure. Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Rogers KA, Thompson PA, Allan JN, Coleman M, Sharman JP, Cheson BD, Jones D, Izumi R, Frigault MM, Quah C, Raman RK, Patel P, Wang MH, Kipps TJ. Phase II study of acalabrutinib in ibrutinib-intolerant patients with relapsed/refractory chronic lymphocytic leukemia. Haematologica. 2021 Sep 1;106(9):2364-2373. doi: 10.3324/haematol.2020.272500. PMID 33730844
- [Derived] Mato AR, Nabhan C, Barr PM, Ujjani CS, Hill BT, Lamanna N, Skarbnik AP, Howlett C, Pu JJ, Sehgal AR, Strelec LE, Vandegrift A, Fitzpatrick DM, Zent CS, Feldman T, Goy A, Claxton DF, Bachow SH, Kaur G, Svoboda J, Nasta SD, Porter D, Landsburg DJ, Schuster SJ, Cheson BD, Kiselev P, Evens AM. Outcomes of CLL patients treated with sequential kinase inhibitor therapy: a real world experience. Blood. 2016 Nov 3;128(18):2199-2205. doi: 10.1182/blood-2016-05-716977. Epub 2016 Sep 6. PMID 27601462
- See also: redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-208&attachmentIdentifier=72dbec9f-2ece-4aea-9063-66b3dde927a3&fileName=ACE-CL-208_CSP_redacted.pdf&versionIdentifier=
- See also: redacted CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-208&attachmentIdentifier=8a1895db-ca33-436f-9813-165266a792f9&fileName=ACE-CL-208_CSR_Synopsis_redacted.pdf&versionIdentifier=
- See also: redacted SAP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=ACE-CL-208&attachmentIdentifier=d7996622-d37e-4abe-81a8-d64bf83aed7b&fileName=ACE-CL-208_SAP_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: For the ACE-CL-208 program, Study Terminated by Sponsor refers to the following: Patients receiving treatment benefits will continue to be provided with study medication in the Post Final Analysis Management of the trial. Sponsor has terminated further data collection for analysis and reporting
Groups:
- Acalabrutinib: Acalabrutinib 100 mg BID
Period: Overall Study
Arm/Group | Acalabrutinib
Started | 60
Completed | 0
Not Completed | 60
Not completed — Death | 13
Not completed — Withdrawal by Subject | 6
Not completed — Active, not recruiting | 40
Not completed — Complicating disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.2 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 38
Race/Ethnicity, Customized [Number; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 54
  Not Reported | 4
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  Native Hawaiian or Other Pacific Islander | 0
  White | 56
  Other | 1
  Not Reported | 2
Region of Enrollment [Number; unit: Participants]
  United States | 49
  Europe | 11

OUTCOME MEASURES:

1. Primary Outcome: The Overall Response Rate (ORR) of ACP-196 (Acalabrutinib)
Description: The overall response rate (ORR) of ACP-196 (acalabrutinib) in subjects with relapsed / refractory CLL who are intolerant of ibrutinib therapy.
  ORR is defined as the proportion of subjects achieving a best overall response (BOR) of either complete remission (CR), complete remission with incomplete bone marrow recovery (CRi), nodular partial remission (nPR), or partial remission (PR) at or before initiation of subsequent anticancer therapy. ORR will be analyzed per investigator's assessment.
Time Frame: From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to approximately 4 years and 7 months). 1 cycle = 28 days
Population: All Treated Population
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Percentage of participants | 70.0 [56.8 to 81.2]

2. Secondary Outcome: Progression-Free Survival
Description: The progression-free survival of ACP-196 (acalabrutinib) in subjects with relapsed / refractory CLL who are intolerant of ibrutinib therapy.
  PFS is calculated as date of disease progression or death (censoring date for censored subjects) - first dose date + 1.
Time Frame: From the date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years).
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Months | NA [33.7 to NA] — not estimable; insufficient number of participants with events

3. Secondary Outcome: Duration of Response
Description: The duration of response of ACP-196 (acalabrutinib) in subjects with relapsed / refractory CLL who are intolerant of ibrutinib therapy.
  DOR is calculated as date of disease progression or death (censoring date for censored subjects) - date of achieving the first CR, CRi, nPR, or PR + 1.
Time Frame: as for outcome 2
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Months | NA [29.9 to NA] — not estimable; insufficient number of participants with events

4. Secondary Outcome: Time-to-Next Treatment
Description: The time to next treatment of ACP-196 (acalabrutinib) in subjects with relapsed / refractory CLL who are intolerant of ibrutinib therapy.
  TTNT is defined as the time from date of first acalabrutinib treatment to date of institution of subsequent anticancer therapy for CLL or death due to any cause, whichever comes first. Subjects who do not have the above specified events prior to the data cutoff date will be censored at the date of last visit. TTNT will be calculated as follows:
  (Earlier date of institution of subsequent anticancer therapy for CLL or date of death due to any cause) - date of first dose + 1. For censored subjects, date of last visit will replace earlier date of use of subsequent anticancer therapy for CLL or date of death due to any cause in the calculation.
Time Frame: From date of the first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years)
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Months | 44.0 [27.4 to NA] — not estimable; insufficient number of participants with events

5. Secondary Outcome: Overall Survival
Description: The overall survival of ACP-319 (acalabrutinib) in subjects with relapsed/refractory CLL who are intolerant of ibrutinib therapy
Time Frame: as for outcome 4
Population: All Treated Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 60
Months | NA [NA to NA] — not estimable; insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From first dose of study drug until 30 days post last dose through study completion. An average of 5 years.
Arm/Group | Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 13/60
Serious Adverse Events (participants affected / at risk) | 32/60
Other Adverse Events (participants affected / at risk) | 60/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Injection site haemorrhage (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (4)
Pyrexia (General disorders) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 7 (8)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 (1)
Pneumonia viral (Infections and infestations) | 1 (1)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Respiratory fume inhalation disorder (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Chronic myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 3 (3)
Confusional state (Psychiatric disorders) | 1 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypertension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=60)
Anaemia (Blood and lymphatic system disorders) | 10 (25)
Eosinophilia (Blood and lymphatic system disorders) | 1 (2)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Lymph node pain (Blood and lymphatic system disorders) | 2 (3)
Lymphocytosis (Blood and lymphatic system disorders) | 4 (5)
Neutropenia (Blood and lymphatic system disorders) | 9 (18)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Polycythaemia (Blood and lymphatic system disorders) | 1 (2)
Spontaneous haemorrhage (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (7)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1)
Cardiorenal syndrome (Cardiac disorders) | 1 (1)
Extrasystoles (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ear discomfort (Ear and labyrinth disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 2 (2)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 4 (4)
Vertigo (Ear and labyrinth disorders) | 3 (3)
Goitre (Endocrine disorders) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Thyroid mass (Endocrine disorders) | 1 (1)
Cataract (Eye disorders) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Ocular hyperaemia (Eye disorders) | 1 (1)
Retinal tear (Eye disorders) | 1 (1)
Retinopathy (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Vitreous floaters (Eye disorders) | 2 (2)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 7 (8)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Barrett's oesophagus (Gastrointestinal disorders) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (12)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 32 (50)
Dry mouth (Gastrointestinal disorders) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Gastric polyps (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Haematochezia (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 2 (2)
Hiatus hernia (Gastrointestinal disorders) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 15 (16)
Oesophagitis (Gastrointestinal disorders) | 1 (1)
Oral blood blister (Gastrointestinal disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 4 (6)
Toothache (Gastrointestinal disorders) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (7)
Asthenia (General disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Chills (General disorders) | 6 (6)
Cyst (General disorders) | 1 (1)
Fatigue (General disorders) | 15 (21)
Feeling cold (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Inflammation (General disorders) | 1 (1)
Influenza like illness (General disorders) | 7 (7)
Localised oedema (General disorders) | 5 (7)
Malaise (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 5 (6)
Oedema (General disorders) | 3 (3)
Oedema peripheral (General disorders) | 10 (12)
Pain (General disorders) | 3 (3)
Peripheral swelling (General disorders) | 3 (3)
Pyrexia (General disorders) | 12 (17)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Portal hypertension (Hepatobiliary disorders) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 2 (2)
Hypogammaglobulinaemia (Immune system disorders) | 2 (2)
Immunodeficiency (Immune system disorders) | 1 (1)
Bronchiolitis (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4)
Cellulitis (Infections and infestations) | 1 (1)
Chronic sinusitis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 3 (5)
Conjunctivitis (Infections and infestations) | 2 (2)
Diverticulitis (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Escherichia bacteraemia (Infections and infestations) | 1 (1)
Folliculitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gingivitis (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Hepatitis b reactivation (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 1 (1)
Infected bite (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (2)
Lower respiratory tract infection (Infections and infestations) | 2 (8)
Nail infection (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Onychomycosis (Infections and infestations) | 1 (1)
Oral fungal infection (Infections and infestations) | 1 (1)
Oral herpes (Infections and infestations) | 2 (3)
Otitis media (Infections and infestations) | 3 (6)
Pneumonia (Infections and infestations) | 8 (13)
Pseudomonas infection (Infections and infestations) | 1 (1)
Pyelitis (Infections and infestations) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1)
Pyuria (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (5)
Rhinitis (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 9 (16)
Skin infection (Infections and infestations) | 3 (3)
Strongyloidiasis (Infections and infestations) | 1 (1)
Tinea infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 20 (34)
Urinary tract infection (Infections and infestations) | 8 (17)
Vulvovaginal mycotic infection (Infections and infestations) | 2 (5)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (3)
Aortic pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 26 (32)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 9 (19)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (3)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Postoperative hypertension (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Scratch (Injury, poisoning and procedural complications) | 1 (1)
Skin abrasion (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 3 (3)
Spinal fracture (Injury, poisoning and procedural complications) | 2 (3)
Subdural haematoma (Injury, poisoning and procedural complications) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (2)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (6)
Anticonvulsant drug level increased (Investigations) | 1 (1)
Blood creatinine increased (Investigations) | 2 (2)
Blood phosphorus decreased (Investigations) | 1 (1)
Cardiac murmur (Investigations) | 2 (2)
Liver function test abnormal (Investigations) | 1 (1)
Liver function test increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (1)
Lymphocyte count increased (Investigations) | 6 (7)
Neutrophil count decreased (Investigations) | 7 (10)
Platelet count decreased (Investigations) | 6 (8)
Prostatic specific antigen increased (Investigations) | 1 (1)
Transaminases increased (Investigations) | 1 (1)
Weight decreased (Investigations) | 4 (7)
Weight increased (Investigations) | 8 (10)
Decreased appetite (Metabolism and nutrition disorders) | 5 (8)
Fluid overload (Metabolism and nutrition disorders) | 1 (1)
Folate deficiency (Metabolism and nutrition disorders) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 4 (4)
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (6)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (13)
Hypophosphataemia (Metabolism and nutrition disorders) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1)
Iron deficiency (Metabolism and nutrition disorders) | 1 (1)
Vitamin d deficiency (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 (17)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (18)
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Diastasis recti abdominis (Musculoskeletal and connective tissue disorders) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 (7)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 (8)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteosclerosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 (9)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (7)
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma of bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Haemangioma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (10)
Tumour flare (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Arachnoid cyst (Nervous system disorders) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 19 (26)
Headache (Nervous system disorders) | 26 (29)
Hypersomnia (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 5 (5)
Lethargy (Nervous system disorders) | 2 (2)
Memory impairment (Nervous system disorders) | 2 (2)
Migraine (Nervous system disorders) | 1 (1)
Migraine with aura (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Sensory loss (Nervous system disorders) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (3)
Tremor (Nervous system disorders) | 4 (4)
Adjustment disorder with depressed mood (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 7 (8)
Insomnia (Psychiatric disorders) | 6 (6)
Nightmare (Psychiatric disorders) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (2)
Chronic kidney disease (Renal and urinary disorders) | 1 (2)
Dysuria (Renal and urinary disorders) | 2 (3)
Glomerulosclerosis (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (9)
Micturition urgency (Renal and urinary disorders) | 2 (2)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Nocturia (Renal and urinary disorders) | 4 (6)
Pollakiuria (Renal and urinary disorders) | 5 (5)
Renal impairment (Renal and urinary disorders) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 3 (3)
Adnexa uteri cyst (Reproductive system and breast disorders) | 1 (1)
Prostatic obstruction (Reproductive system and breast disorders) | 1 (1)
Spermatocele (Reproductive system and breast disorders) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (25)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 9 (11)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Blood blister (Skin and subcutaneous tissue disorders) | 1 (1)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Ecchymosis (Skin and subcutaneous tissue disorders) | 5 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (8)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1)
Ingrown hair (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 8 (11)
Onychoclasis (Skin and subcutaneous tissue disorders) | 2 (2)
Petechiae (Skin and subcutaneous tissue disorders) | 5 (6)
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (7)
Purpura (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 12 (13)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (5)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 7 (8)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1)
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 1 (1)
Aortic stenosis (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 8 (10)
Hypotension (Vascular disorders) | 5 (5)
Intermittent claudication (Vascular disorders) | 1 (1)
Lymphoedema (Vascular disorders) | 2 (3)
Peripheral coldness (Vascular disorders) | 1 (1)
Thrombophlebitis superficial (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2020-06-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT02717611/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/11/NCT02717611/SAP_001.pdf